CLINICAL TRIAL: NCT00211575
Title: Clinical Utility of an Instrument in the Evaluation of Young Children With Suspected Asthma
Brief Title: Instrument Utility for Suspected Asthma (0000-042)(COMPLETED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-042; 042; 2005_073
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
This research study was designed to help improve the diagnosis and treatment of asthma in young children. An interventional strategy using a scoring system based on risk factors and symptoms/episodes was tested to determine its ability to identify children likely to benefit from induction of asthma controller therapy at an early age. The score was derived through completion of a survey instrument referred to as the asthma risk questionnaire (ARQ). The utility of the ARQ along with the health care utilization and use of controller therapy for respiratory illnesses within one year were examined.

ELIGIBILITY:
Inclusion Criteria:

* Children less than or equal to 6 years of age who had at least 1 year prior episode of wheezing

Exclusion Criteria:

* Children with other systemic or chronic respiratory disease and children who used an asthma controller medication with the 6 weeks prior to enrollment

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Utility of ARQ as measured by the percentage of children started on any asthma medication and characteristics of those diagnosed with asthma

SECONDARY OUTCOMES:
Percentage of children with recurrent wheezing, placed on controller therapy, number of steroid courses and need for urgent medical care at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC